CLINICAL TRIAL: NCT01717053
Title: A Phase II Trial of Abiraterone Acetate, Radiotherapy and Short-Term Androgen Deprivation in Men With Unfavorable Risk Localized Prostate Cancer
Brief Title: Abiraterone, Radiotherapy and Short-Term Androgen Deprivation in Unfavorable Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00044071
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Radiotherapy; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): Abiraterone Acetate, Radiotherapy and Short Term Androgen Deprivation. Prednisone will be prescribed concurrently with Abiraterone acetate.
  Interventions: Drug: Abiraterone acetate; Drug: Androgen deprivation; Radiation: Radiation Therapy; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — 1000 mg orally once a day for 6 months.
  Other Names: Zytiga
Drug: Androgen deprivation — LHRH analog (at discretion of treating physician) will be administered over 6 months (for example, leuprolide acetate 22.5mg IM or goserelin acetate 10.8mg SC given every 3 months for 2 doses).
Radiation: Radiation Therapy — Daily (Monday-Friday) for 8 weeks, final dose of 75-80 Gy
Drug: Prednisone — 5 mg tablet once daily for 6 months.

SUMMARY:
The addition of abiraterone acetate to standard treatment of radiotherapy and short-term androgen deprivation will increase the frequency of undetectable PSA.

DETAILED DESCRIPTION:
This is a single arm two-site study of 37 men with unfavorable prostate cancer (defined as having a single high risk factor). Patients will concurrently initiate 6 months of standard-of-care GNRH agonist therapy and once daily abiraterone acetate/prednisone. After 2 months of lead-in hormonal treatment, definitive standard-of-care prostate/seminal vesicle radiotherapy will be delivered, to a total dose of 75-80 Gy.

ELIGIBILITY:
Inclusion Criteria:

* One of the following high risk criteria:
* Gleason Score 7 with PSA ≤ 20 ng/ml and clinical T1-2, or
* Gleason Score 8-10, PSA ≤ 20 ng/ml and clinical T1-2a, or
* PSA 10.1-40 ng/ml with GS < 7 and clinical T1-2, or
* Clinical T3 with Gleason Score < 7 and PSA ≤ 10 ng/ml.
* ECOG Performance Status ≤ 1
* Digital rectal exam within 90 days of registration on study
* CBC with differential with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3, Platelets > 100,000/µL and Hemoglobin ≥ 9g/dL
* Serum potassium ≥ 3.5 mEq/L
* Serum albumin > 3.0 g/dl
* Total bilirubin < 1.5 X of institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) < 1.5 X ULN
* Calculated creatinine clearance > 60 mL/min
* Age > 18 years
* Able to swallow a whole tablet and take abiraterone acetate on an empty stomach (defined as no food for two hours before and one hour after abiraterone acetate ingestion)
* Ability to understand and sign a written informed consent document
* Written authorization for use and release of health and research study information has been obtained
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Subjects who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protections as determined acceptable by the principal investigator during the study and for 1 week after the last dose of abiraterone acetate.

Exclusion Criteria:

* Bone, visceral or soft tissue metastasis, including lymph nodes (>2 cm in longest diameter)
* Prior therapy for prostate cancer [Exceptions: LHRH agonist or antagonist may have been initiated within 30 days prior to enrollment. Bicalutamide may have been given within 60 days of enrollment as long as it has been stopped at least 7 days before enrollment and total duration was no longer than 30 days. This is to allow enrollment of those who have been given bicalutamide as a bridge for LHRH agonist/antagonist. It is highly unlikely a short non-overlapping course of bicalutamide will interact with abiraterone acetate in a measurable way. Previous alpha-reductase inhibitor use allowed IF patient has not been taking for at least 30 days prior to abiraterone acetate initiation, OR if alpha reductase inhibitor was not used as a primary treatment of prostate cancer and the PSA on alpha-reductase inhibitor remains within eligibility when doubled. ]
* Known serum testosterone ≤ 150 ng/dl or symptoms of hypogonadism (fatigue, hot flashes, hair loss, loss of muscle mass, osteoporosis, low libido, depression) prior to ADT initiation not explained by other medical co-morbidity OR history of testosterone supplement. If questionable, serum testosterone level greater than 150 ng/dl can be used to exclude hypogonadism.
* Previous malignancy within 3 years other than non-melanomatous skin cancer and non-muscle invasive bladder cancer
* Previous pelvic radiotherapy that would prevent prostate/SV irradiation
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
* History of gastrointestinal disorders that may interfere with the absorption of study drug (including gastric bypass surgery)
* Concurrent spironolactone use
* Significant concurrent medical condition that would make prednisone/prednisolone use contraindicated or would interfere with the patient's ability to participate in the trial
* Receiving any investigational agents currently or within 30 days prior to study screening
* Prior demonstrated hypersensitivity, intolerance or allergy to abiraterone acetate, prednisone or their excipients
* Active co-morbidity, defined as follows:

  * Chronic liver disease with cirrhosis (Child-Pugh B or C) or active hepatitis B or C
  * History of pituitary or adrenal dysfunction
  * Poorly controlled diabetes mellitus (A1c >9% or history of complications including peripheral neuropathy, end organ damage, hospitalization, amputation)
  * Poorly controlled glaucoma
  * Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III-IV heart disease or known cardiac ejection fraction measurement of < 50% at baseline.
  * Clinical evidence of active infection of any type, including active or symptomatic viral hepatitis.
  * Known immune deficiency and/or HIV-positive patients
  * Any medical condition that warrants long-term corticosteroid use in excess of study dose
* Patients taking strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital)
* Any condition that in the opinion of the Principal Investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing the study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Koontz BF, Hoffman KE, Halabi S, Healy P, Anand M, George DJ, Harrison MR, Zhang T, Berry WR, Corn PG, Lee WR, Armstrong AJ. Combination of Radiation Therapy and Short-Term Androgen Blockade With Abiraterone Acetate Plus Prednisone for Men With High- and Intermediate-Risk Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1271-1278. doi: 10.1016/j.ijrobp.2020.11.059. Epub 2020 Nov 28. PMID 33259932

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone+Radiotherapy+ADT: Abiraterone Acetate, Radiotherapy and Short Term Androgen Deprivation. Prednisone will be prescribed concurrently with Abiraterone acetate.
Period: Overall Study
Arm/Group | Abiraterone+Radiotherapy+ADT
Started | 37
Completed | 33
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Undetectable PSA (Prostate-Specific Antigen) at 1 Year
Description: The percentage of patients with undetectable PSA after 1 year will be calculated. Undetectable PSA is defined as a measurement of <0.1 ng/mL.
Time Frame: 1 year
Population: This analysis includes all patients that completed protocol therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 33
percentage of participants | 54.54

2. Secondary Outcome: Time to PSA Nadir
Description: The median time in months to the lowest PSA value from the start of study therapy.
Time Frame: 1 year
Population: This analysis includes all patients that completed protocol therapy.
Measure: Median (Full Range); unit: months
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 33
months | 8.9 [2.9 to 39.3]

3. Secondary Outcome: PSA Nadir Value
Description: The lowest PSA value from the start of study therapy.
Time Frame: 1 year, 2 years
Population: This analysis includes all patients that completed protocol therapy.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 33
ng/mL
  Year 1 | 0.03 [0 to 0.44]
  Year 2 | 0.03 [0 to 0.36]

4. Secondary Outcome: Percentage of Participants With Biochemical Progression-free Survival (BPFS)
Description: Disease progression defined as Phoenix RTOG definition of nadir PSA + 2ng/ml or initiation of salvage therapy not imaging. The two outcomes use different measures (biochemical as measured by PSA increase vs radiographic as measured by imaging), yielding different results in this case.
Time Frame: 36 and 48 months
Population: Men with unfavorable prostate cancer (defined as having a single high risk factor)
Measure: Number; unit: percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 33
percentage of participants
  36 months | 96.96
  48 months | 96.96

5. Secondary Outcome: Metastasis or Systemic Therapy
Description: Time to either imaging indicating metastasis or beginning a new systemic therapy. This is a distinctly different measure from number 4 above. The two outcomes use different measures (biochemical as measured by PSA increase vs radiographic as measured by imaging), yielding different results in this case.
Time Frame: up to 5 years (60 months)
Population: Men with unfavorable prostate cancer (defined ad having a single high risk factor)
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 33
months | 60 [NA to NA] — Insufficient number of participants with events.

6. Secondary Outcome: Testosterone Recovery
Description: Time to testosterone recovery
Time Frame: up to 5 years
Population: Men with unfavorable prostate cancer (defined ad having a single high risk factor)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 37
months | 9.2 [9 to 12.3]

7. Secondary Outcome: PSA < 1.5ng/ml in Setting of Non-castrate Testosterone
Description: Percentage of men with 1, 2, 3, 4 and 5 year PSA < 1.5ng/ml in setting of non-castrate testosterone.
Time Frame: 1 year, 2 years, 3 years, 4 years, 5 years
Population: Men with unfavorable prostate cancer (defined as having a single high risk factor)
Measure: Number; unit: percentage of patients
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 33
percentage of patients
  1 year | 100
  2 years | 100
  3 years | 90.91
  4 years | 90.91
  5 years | 90.91

8. Secondary Outcome: Safety and Tolerability
Description: The number of patients experiencing an adverse event of at least grade 3 that is possibly, probably, or definitely related to study therapy per CTCAE version 4.0.
Time Frame: 6 months
Population: This analysis includes all patients that completed protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone+Radiotherapy+ADT
Number analyzed (Participants) | 33
Participants | 12

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Abiraterone+Radiotherapy+ADT
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 4/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone+Radiotherapy+ADT (N=37)
Fever (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Other, specify: Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone+Radiotherapy+ADT (N=37)
Anemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify: Irregular heart beats (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify: ""slight off balance and fluid in ears"" (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify: Slight off balance (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify: Left eye ""stye with morning crustiness"" (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Esophageal pain (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Bowel urgency (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Guaiac positive stools (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Intermittent ""mucous loose stool"" (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Pt reports intermittent frank red blood on stool (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: diverticulitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: intermittent rectal bleeding (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: urgency with bowels (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 24
General disorders and administration site conditions - Other, specify: Injury left hand (General disorders) | 1
General disorders and administration site conditions - Other, specify: Occasional cramping (General disorders) | 1
General disorders and administration site conditions - Other, specify: Perineal pain (General disorders) | 1
Injection site reaction (General disorders) | 1
Irritability (General disorders) | 3
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Infections and infestations - Other, specify: C diff colitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Burn (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify:Chigger bite (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify: Injury to Right Shin (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify: face injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 12
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 1
Investigations - Other, specify: Blood Urea Nitrogen 20(7-18); 20 (8-20) (Investigations) | 1
Investigations - Other, specify: Blood Urea Nitrogen 21 (8-20) (Investigations) | 1
Investigations - Other, specify: Blood Urea Nitrogen 23 (7-18); 20 (8-20) (Investigations) | 1
Investigations - Other, specify: Blood urea nitrogen 28;18 (Investigations) | 1
Investigations - Other, specify: CO2 level (carbon dioxide) 31 (Investigations) | 1
Investigations - Other, specify: CO2 level (carbon dioxide)31 (Investigations) | 1
Investigations - Other, specify: CO2 level (carbon dioxide)31 (23-30) (Investigations) | 1
Investigations - Other, specify: Decreased ALT, <12 (7-56) (Investigations) | 1
Investigations - Other, specify: Elevated CO2 (Carbon Dioxide) level at 31 (23-30) (Investigations) | 1
Investigations - Other, specify: Elevated Total Bilirubin (Investigations) | 1
Investigations - Other, specify: Elevated Total Bilirubin, decreased at 1.5 (Investigations) | 1
Investigations - Other, specify: Increased Albumin 5.0 (3.5-4.7) (Investigations) | 1
Investigations - Other, specify: Increased CO2 (carbon dioxide) level, 31 (Investigations) | 1
Investigations - Other, specify: Low Chloride 96 (98-108) (Investigations) | 1
Investigations - Other, specify: Low Chloride 97;on 3/31- 96 (98-108) (Investigations) | 1
Investigations - Other, specify: Low serum creatinine, 0.66 (Investigations) | 1
Investigations - Other, specify: Minimally increased @ 32 (23-30) (Investigations) | 1
Investigations - Other, specify: Serum Carbon Dioxide Level 32;28 (23-30) (Investigations) | 1
Investigations - Other, specify: Serum Carbon Dioxide Level 34;29 (23-30) (Investigations) | 1
Investigations - Other, specify: Weight loss, 83.7 kg (88 kg on 6/4/15) (Investigations) | 1
Platelet count decreased (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 3
Metabolism and nutrition disorders - Other, specify: Possible mineralcorticoid excess (hypokalemia) (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: elevated ALT/AST (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: low Total Protein level- 5.8 (6.1-8.1) (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Chronic left hip/sciatica pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Decreased strength & endurance (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: L4-L5 procedure on 8/4/15 (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Right Lower Extremity leg spasm (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Right flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: bursitis, left knee (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: restless legs (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify: Chronic sciatic back pain (Nervous system disorders) | 1
Nervous system disorders - Other, specify: Pre-treatment, chronic sciatic back pain (Nervous system disorders) | 1
Nervous system disorders - Other, specify: lightheaded, when standing (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 5
Libido decreased (Psychiatric disorders) | 6
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify: Dysuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Increased urination (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Nocturia (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify: Slow urinary stream (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Urinary hesistancy (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Urinary hesitancy (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, specify: Weak urinary stream (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: nocturia (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: weak stream (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 20
Urinary incontinence (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 6
Urinary urgency (Renal and urinary disorders) | 5
Erectile dysfunction (Reproductive system and breast disorders) | 3
Gynecomastia (Reproductive system and breast disorders) | 2
Perineal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify: Dry nose (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify: (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Basal cell carcinoma of left ear (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Melanoma of lower back (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Melanoma of right shoulder (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Soft non-tender area on lower leg (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: skin pallor, pale (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 28
Hypertension (Vascular disorders) | 22
Vascular disorders - Other, specify: Facial petechiae ""from force of vomiting"" per pt (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT01717053/Prot_SAP_000.pdf